CLINICAL TRIAL: NCT06230367
Title: Harnessing the Power of Text Messaging to Reduce HIV Incidence in Adolescent Males Across the United States
Brief Title: Sexual Health Advocacy for Guys - a Text Messaging-based HIV Prevention Program for Guys Who Are Into Guys
Acronym: SHAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01HD108738 (NIH)
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention or control group
Who Masked: Participant
Masking Description: Control group content is written to affect an experience as if one were in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHAG (Sexual Health Advocacy for Guys) (Experimental): Young people assigned to the intervention arm will receive ~9 weeks of daily text messages that talk about healthy sexuality and ways to reduce HIV risk. After a 3 month 'quiet' period, they will receive a week of review messages. Messages are based upon the information-motivation-behavioral model of preventive behavior.
  Interventions: Behavioral: Sexual health advocacy for guys
- Attention-matched control (Placebo Comparator): Young people assigned to the control arm will receive ~9 weeks of daily text messages that talk about healthy lifestyle, such as self-esteem and physical exercise. After a 3 month 'quiet' period, they will receive a week of review messages.
  Interventions: Behavioral: Healthy lifestyle control

INTERVENTIONS:
Behavioral: Sexual health advocacy for guys — 5 month HIV prevention program delivered via text messaging
  Arms: SHAG (Sexual Health Advocacy for Guys)
Behavioral: Healthy lifestyle control — 5 month control group program delivered via text messaging
  Arms: Attention-matched control

SUMMARY:
SHAG is a text messaging-based HIV prevention program designed for cisgender sexual minority boys and men 13-20 years of age across the United States. Investigators will test it against a control group that receives messages about healthy lifestyle.

DETAILED DESCRIPTION:
SHAG is a text messaging-based HIV prevention program designed for cisgender sexual minority boys and men 13-20 years of age across the United States. Investigators will test it against a control group that receives messages about healthy lifestyle. Harnessing the power of technology, young people will be recruited online and largely enrolled digitally. The main outcome of interest is HIV incidence. The impact of the intervention on STI testing and pre-exposure prophylaxis (PrEP) will also be examined.

ELIGIBILITY:
Inclusion Criteria:

1. have been assigned male sex at birth and currently have a cisgender identity;
2. be aged 13-22 years old;
3. have had anal sex in the past 12 months;
4. be English-speaking;
5. exclusively own a cell phone with an unlimited text messaging plan and intend to have the same cell phone number for the next 6 months;
6. have Internet access to complete online surveys;
7. provide informed assent for those under 18, and consent for those 18 years of age and older, including a capacity to consent and a positive self-safety assessment;
8. Willing to take an OraQuick home test to confirm HIV negativity for youth who are 19-20 years of age or 18 years old and graduated high school. If they agree to do the test but do not upload a photo of their result, they will be eligible if they self-report a negative sero-status. Youth 18 years old who have not graduated high school, and 13-17 years of age will be asked to take a home test. If they determine that they cannot do so safely, they will be allowed to self-report their sero-status; and
9. not currently enrolled in another HIV prevention program; or
10. know anyone already enrolled in the RCT.

Exclusion Criteria:

* Being HIV positive

Ages: 13 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
HIV Incidence | 12-months post-intervention and immediately post-intervention
  HIV Incidence determined by home testing kit

SECONDARY OUTCOMES:
Self-reported HIV incidence | Post-Intervention, 3-months post, 6-months post, 9-months post, 12-month post
  Self-reported HIV Status
Proportion of Participants Testing for an STI | 12-month post intervention and immediately post-intervention
  This outcome will be measured as a cumulative indicator of whether the individual has tested for an STI
Proportion of Participants having used PrEP/PEP | 12-month post-Intervention and immediately post-intervention
  This outcome will be measured as a cumulative indicator of whether the individual has used pre-exposure or post-exposure prophylaxis for HIV

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovative Public Health Research, San Clemente, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level de-identified data will be made available through controlled access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available starting 12 months after the grant ends.
Access Criteria: * Data access requires sponsorship by an Institution on behalf of the prospective recipient.
  * Requester must provide documentation of local IRB approval
  * Requester agrees to make results of studies using the data available to the larger scientific community
  * Requester must provide a letter of collaboration with the primary study investigator
  * Use of the data is limited to not-for-profit organizations
  * Use of the data is limited to health purposes

REFERENCES:
- [Derived] Ybarra ML, Feaster DJ, Garofalo R, Bull S. Sexual Health Advocacy for Guys (SHAG): a randomized trial of the impact of a text-messaging program on HIV incidence and STI testing among a national sample of sexual minority cisgender adolescent and young adult men. Trials. 2025 Jan 6;26(1):9. doi: 10.1186/s13063-024-08540-9. PMID 39762976